CLINICAL TRIAL: NCT01194050
Title: Erlotinib (Tarceva) in Routine Clinical Practice for First Line Maintenance Therapy (1LM) in Patients With Advanced Non Small Cell Lung Cancer (NSCLC)
Brief Title: An Observational Study of Tarceva (Erlotinib) in Routine Practice For First Line Maintenance Therapy in Patients With Non Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22816
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will investigate the tolerability and efficacy of Tarceva (erlotinib) in daily clinical practice under routine conditions in patients with locally advanced or metastatic non small cell lung cancer. Data will be collected for approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with locally advanced or metastatic non-small cell lung cancer (stage IIIb or IV) with stable disease after 4 cycles of standard platinum-based first-line chemotherapy

Exclusion Criteria:

* Not willing or not able to sign written informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non small cell lung cancer patients
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Overall survival at 1 year | 12 months

SECONDARY OUTCOMES:
Tolerability of Tarceva in daily clinical practice under routine conditions | 12 months
Efficacy of Tarceva in daily clinical practice under routine conditions | 12 months
Reproducibility of the results of the controlled SATURN study | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Villingen-Schwenningen, Germany